CLINICAL TRIAL: NCT06193109
Title: The Prognostic Impact of Right Ventricular Systolic Dysfunction on the Survival of Patients With Sepsis and Septic Shock
Status: Completed | Type: Observational
Sponsor: Burapha University (Other)
Responsible Party: Principal Investigator, Sukrisd Koowattanatianchai, Assistant Professor Dr., Burapha University
Other Study IDs: Burapha university
Record Dates: First submitted 2023-12-12; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Sepsis and Septic Shock
Keywords: right ventricular systolic dysfunction
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the patients with sepsis or septic shock: devide two groups : (1) They had right ventricular dysfunction and (2) They had no right venticular dysfunction.

INTERVENTIONS:
Other:  — the patients with sepsis and septic shock were performed echocardiography for detecting right ventricular systolic function

SUMMARY:
This study sought to evaluate the association of right ventricular systolic dysfunction and 28-day in-hospital mortality in patients with sepsis and septic shock. Prospective cohort study of adult patients admitted at Burapha university hospital from October 1, 2022 through June 30, 2023 for sepsis and septic shock, who had an echocardiogram within 72 hours after admission for evaluating right ventricular systolic function. Right ventricular systolic dysfunction was defned by the American Society of Echocardiography criteria. Outcomes included 28-day in-hospital mortality, maximal blood lactate, length of intensive care unit(ICU) stay and duration of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* diagnosed with sepsis or septic shock according to Sepsis-3 criteria
* received an echocardiogram within 72 hours after admission

Exclusion Criteria:

* prior diagnosis of pulmonary hypertension,
* cor-pulmonale,
* significant valvular heart disease,
* acute coronary syndrome,
* aortic dissection,
* heart failure
* inability to follow up within 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective study was conducted at Burapha University Hospital, enrolling admitted patients diagnosed with sepsis and septic shock. Echocardiography was performed on these patients within 72 hours after admission
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
28 days in-hospital mortality | October 1, 2022 and June 30, 2023
  28 days in hospital mortality in patients with sepsis or septic shock

SECONDARY OUTCOMES:
The prevalence of right ventricular systolic dysfunction | October 1, 2022 and June 30, 2023
  The prevalence of right ventricular systolic dysfunction in patients with sepsis and septic shock
Blood lactate levels | October 1, 2022 and June 30, 2023
  Blood lactate levels in patients with sepsis and septic shock
Lenght of ICU stay | October 1, 2022 and June 30, 2023
  Lenght of ICU stay in patients with sepsis and septic shock
Duration of mechanical ventilation | October 1, 2022 and June 30, 2023
  Duration of mechanical ventilation in patients with sepsis and septic shock

CONTACTS AND LOCATIONS:
Locations (1):
- Burapha University Hospital, Muang Chonburi, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after finishing the research and for 1 year after submission

REFERENCES:
- [Derived] Koowattanatianchai S, Kochaiyapatana P, Eungsuwat N, Rangsrisaeneepitak V, Thammakumpee K, Kaladee K. Significance of Right Ventricular Dysfunction in Predicting Short-Term Survival Among Patients With Sepsis and Septic Shock: A Prognostic Analysis. Crit Care Res Pract. 2025 Mar 14;2025:5511135. doi: 10.1155/ccrp/5511135. eCollection 2025. PMID 40125344